CLINICAL TRIAL: NCT07329738
Title: A 3D-Printed Prosthesis Portable Station: The Vancouver Limbkit Project
Brief Title: Single-Subject Research Design on 3D-Printed Prosthetic Sockets
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, William C. Miller, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H22-03708; F22-05611 (Other Grant/Funding Number: The Amputee Coalition of Canada); F24-00369 (Other Grant/Funding Number: War Amps)
Record Dates: First submitted 2025-12-09; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Transtibial Amputees

STUDY DESIGN:
Intervention Model Description: Single-subject design (AB): therefore, each participant goes through two phases:
  A= use regular prosthesis B= use 3D-printed prosthesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (one arm only) (Other): Single-subject design (AB): therefore, each participant goes through two phases:
  A= use regular prosthesis B= use 3D-printed prosthesis
  Interventions: Device: 3D printed prosthetic sockets

INTERVENTIONS:
Device: 3D printed prosthetic sockets — The sockets are 3D printed using Polyethylene Terephthalate Glycol (PETG) filament. The printer used for this process is the Fused Deposition Modelling (Creality Ender 6), equipped with a 1.0 mm nozzle diameter, a print speed of 45mm/s, and a layer thickness of 2 mm. To enhance their strength, the sockets are reinforced with Delta-Lite® plus cast tapes and assembled using a distal push-lock mechanism and plate. The number of reinforcement wraps of the Delta-Lite® differs for each region of the socket. Below the sockets, the same prosthetic components from the previous prosthesis are utilized where possible. Participants wear their 3D printed sockets for an adjustment period (3-7 days) and then come in for a follow-up session to ensure the 3D socket still fits well after their limb has settled into the new system. Once both the prosthetist and participant are happy with the fit, Phase B testing is scheduled.

SUMMARY:
The goal of this single-subject research design (clinical trial) is to assess the functionality of the 3D printed prostheses and to compare them to the existing prostheses in terms of mobility, balance, utility, and comfort. Participants who have a unilateral or bilateral transtibial amputation wear their existing prosthesis for roughly 3 weeks, followed by 3 weeks wearing a 3D printed prosthesis. The research assistants collect data throughout each period remotely, with the exception of one in-person visit to participants' homes to prepare the setting for the virtual evaluation sessions.

DETAILED DESCRIPTION:
Once a participant is recruited and consent is obtained, Phase (A) begins with the research assistants conducting one home visit with the participant. This visit sets up the performance-based outcome measures, provides instructions for performing the tests, explains how to complete the online surveys, and clarifies how to take the video recordings. The research assistants distribute the Sociodemographic and Clinical Characteristics questionnaire to the participant via the UBC Qualtrics platform.

During Phase (A), the participant wears their definitive prosthesis and is remotely evaluated up to three times per week for three weeks. At the end of Phase (A), the participant receives an online self-reported survey to measure the utility of using the definitive prosthesis.

The participant then attends their prosthetic clinic to have measurements and a scan of their residual limb taken for the 3D printed prosthesis. The prosthetists use the "Comb" mobile scanner application, and the scans of the participants are securely stored and de-identified to maintain the confidentiality of the participants' information through the HIPAA-compliant Comb portal. The research assistant prints the prosthesis, which includes implanting a thermal sensor into the prosthesis to monitor the wear time. The participant visits the prosthetic clinic a second time to have the 3D printed prosthesis fitted by the relevant prosthetist in the team. The prosthetist ensures the new prosthesis is properly fitted and appropriate for use before allowing the participant to go home with it.

In Phase (B), the participant uses the 3D-printed prosthesis for three weeks and conducts the same outcome measures. At the end of Phase (B), the participant receives an online self-reported survey to measure the utility of using the 3D printed prosthesis.

Participants drop off the 3D-printed prostheses at their prosthetic clinics at the end of the study. Then the RA collects all the 3D printed prostheses to keep them in a locked cabinet in the principal investigator's office at the University of British Columbia.

The participant then has a one-to-one virtual semi-structured interview to explore their experiences with the 3D printed prosthesis.

A separate focus group is conducted with prosthetists involved in this study to obtain their feedback and suggestions regarding the Limbkit.

ELIGIBILITY:
Inclusion Criteria:

* are adults 19+ years,
* have a unilateral or bilateral transtibial amputation,
* have an existing definitive prosthesis,
* use their definitive prosthesis two or more consecutive hours per day,
* have no wounds on the residual limb.

Exclusion Criteria:

* are unable to adequately complete self-report measures or communicate well enough to participate in the end of project interview,
* have bilateral upper extremity amputations,
* have poorly controlled comorbidities (e.g., unstable diabetes, advanced heart problems)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test (TUG) | Measurements are collected three times a week for three weeks (nine times) in phase A and three times a week for three weeks (nine times) in phase B.
  Participants rise from a chair, walk three meters, turn around a cone, return to the chair, and sit; time is recorded from start (standing) to finish (sitting). The TUG score is the average of two timed trials.

SECONDARY OUTCOMES:
Four Square Step Test (FSST) | Measurements are collected three times a week for three weeks (nine times) in phase A and three times a week for three weeks (nine times) in phase B.
  Multi-directional stepping through four square positions (sequence: 1→2→3→4→1→4→3→2→1); time is recorded from initial stance in square one until returning to square one. The FSST score is the average of two timed trials.
Activities-Specific Balance Confidence Scale (ABC) | Measurements are collected three times a week for three weeks (nine times) in phase A and three times a week for three weeks (nine times) in phase B.
  A 16-item questionnaire that assesses confidence in avoiding balance loss across daily activities (e.g., walking on an icy sidewalk). Scores range from 0%-100%, with higher scores indicating greater confidence. The ABC score is the average of the 16 items.
Socket comfort was measured with the Socket Comfort Score (SCS) | Measurements are collected three times a week for three weeks (nine times) in phase A and three times a week for three weeks (nine times) in phase B.
  A single-item measure adapted from pain scales in which 0 = extreme discomfort and 10 = optimal comfort.

OTHER OUTCOMES:
Prosthesis evaluation questionnaire (PEQ) | Measurements are collected three times a week for three weeks (nine times) in phase A and three times a week for three weeks (nine times) in phase B. Utility scale measurements are taken twice; once at the end of phase A and again at the end of phase B.
  The questions in the self-report survey (mobility, pain, and utility) are adopted from the well-developed questionnaire, Prosthesis Evaluation Questionnaire (PEQ), for people with lower limb amputation.
  The mobility scale: scores range from 0 to 100, with higher scores indicating better mobility.
  The pain questions include (intensity and frequency) items:
  The pain intensity scores range from 0 to 100. Higher scores indicate less intense pain.
  The pain frequency scores range from 0 to 6, where 0 means "never" and 6 means "all the time" or "almost all the time." Higher scores indicate more frequent pain.
  The utility scale: scores range from 0 to 100, with higher scores indicating better prosthesis utility
Short Physical Performance Battery (SPPB) | Measurements are collected three times a week for three weeks (nine times) in phase A and three times a week for three weeks (nine times) in phase B.
  SPPB includes static standing balance in three postures for 10 seconds, lower limb strength of getting up and sitting on a chair without using the arms, and walking speed at a normal pace. Component scores are summed to produce a total score ranging from 0 to 12. Higher total scores indicate better lower-extremity function/physical performance.
Figure of Eight Walk Test (F8WT) | Measurements are collected three times a week for three weeks (nine times) in phase A and three times a week for three weeks (nine times) in phase B.
  This test requires participants to walk a figure-of-8 around two cones placed 1.5 m apart. The F8WT score is the average of two-timed trials.

CONTACTS AND LOCATIONS:
Overall Officials: William C. Miller, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No